CLINICAL TRIAL: NCT05696379
Title: Angiography Derived Index of Microcirculatory Resistance in Patients With Acute Myocardial Infarction
Status: Completed | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Shengjing Hospital (Other); RenJi Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-0878
Record Dates: First submitted 2022-12-13; First posted 2023-01-25 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2022-12

CONDITIONS: Acute Myocardial Infarction (AMI)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- STEMI with high Angio-IMR: Patients with ST segment elevation myocardial infarction and high Angio-IMR
  Interventions: Other: Angiography derived index of micro-circulatory resistance (Angio-IMR)
- STEMI with low Angio-IMR: Patients with ST segment elevation myocardial infarction and low Angio-IMR
  Interventions: Other: Angiography derived index of micro-circulatory resistance (Angio-IMR)
- NSTEMI with high Angio-IMR: Patients with non-ST segment elevation myocardial infarction and high Angio-IMR
  Interventions: Other: Angiography derived index of micro-circulatory resistance (Angio-IMR)
- NSTEMI with low Angio-IMR: Patients with non-ST segment elevation myocardial infarction and low Angio-IMR
  Interventions: Other: Angiography derived index of micro-circulatory resistance (Angio-IMR)

INTERVENTIONS:
Other: Angiography derived index of micro-circulatory resistance (Angio-IMR) — Angiography derived index of micro-circulatory resistance (Angio-IMR) post percutaneous coronary intervention.

SUMMARY:
Coronary microcirculatory dysfunction has been known to be prevalent even after successful revascularization of acute myocardial infarction (AMI) patients, and has been shown to be associated with poor prognosis. Angiography derived index of micro-circulatory resistance (Angio-IMR) is a novel pressure-wire free approach to assess coronary microvascular disease with great diagnostic performance. The current study will further investigate the prognostic value of Angio-IMR in patients with AMI in multicenter retrospective cohort.

ELIGIBILITY:
Inclusion Criteria:

* Acute myocardial infarction patients who underwent successful percutaneous coronary intervention

Exclusion Criteria:

* No appropriate coronary angiography images (inferior image quality, image loss, severe arteries overlap, or significant artifact)
* Previous coronary artery bypass graft

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted with a diagnosis of acute myocardial infarction underwent successful percutaneous coronary intervention.
Sampling Method: Probability Sample
Enrollment: 5000 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Cardiac death or readmission for heart failure in 1 month | 1 month
  Incidence of cardiac death or readmission for heart failure during first 1 month follow-up.
Cardiac death or readmission for heart failure in 6 months | 6 month
  Incidence of cardiac death or readmission for heart failure during first 6 months follow-up.
Cardiac death or readmission for heart failure in 1 year | 1 year
  Incidence of cardiac death or readmission for heart failure during first 1 year follow-up.
Cardiac death or readmission for heart failure in 2 years | 2 year
  Incidence of cardiac death or readmission for heart failure during first 2 years follow-up.

CONTACTS AND LOCATIONS:
Locations (1):
- Second Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chen Z, Zhang Y, Fang J, Zheng Y, Chen D, Yidilisi A, Zhang X, Liu C, Huang J, Ji R, Chen J, Chen G, Lin P, Hu Y, Xiang J, Wang J, Jiang J. Thorough Physiological Assessment in Non-Culprit Vessels of Patients with Acute Myocardial Infarction: Is It a Required Action? Cardiovasc Drugs Ther. 2025 Sep 6. doi: 10.1007/s10557-025-07768-0. Online ahead of print. PMID 40913743
- [Derived] Chen D, Zhang Y, Yidilisi A, Hu D, Zheng Y, Fang J, Gong Q, Huang J, Dong Q, Pu J, Niu T, Xiang J, Wang J, Jiang J. Combined risk estimates of diabetes and coronary angiography-derived index of microcirculatory resistance in patients with non-ST elevation myocardial infarction. Cardiovasc Diabetol. 2024 Aug 16;23(1):300. doi: 10.1186/s12933-024-02400-1. PMID 39152477
- [Derived] Zhang Y, Pu J, Niu T, Fang J, Chen D, Yidilisi A, Zheng Y, Lu J, Hu Y, Koo BK, Xiang J, Wang J, Jiang J. Prognostic Value of Coronary Angiography-Derived Index of Microcirculatory Resistance in Non-ST-Segment Elevation Myocardial Infarction Patients. JACC Cardiovasc Interv. 2024 Aug 26;17(16):1874-1886. doi: 10.1016/j.jcin.2024.04.048. Epub 2024 Aug 7. PMID 39115479